CLINICAL TRIAL: NCT05406700
Title: A Phase 0 Clinical Trial to Evaluate Drug Concentrations and Pharmacodynamic Parameters of Niraparib in Tumor Tissue of Patients With Surgically Accessible Recurrent IDH 1/2 Gliomas
Brief Title: Niraparib In Recurrent IDH 1/2 Gliomas
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Isabel Arrillaga-Romany, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-762
Record Dates: First submitted 2022-04-25; First posted 2022-06-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Low-grade Glioma; IDH2 Gene Mutation; Recurrent Glioma; IDH1 Mutation; Glioma, Malignant
Keywords: Low-grade Glioma; IDH2 Gene Mutation; Recurrent Glioma; IDH1 Mutation; Glioma, Malignant
MeSH Terms: conditions — Glioma | interventions — niraparib; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A Treatment with Niraparib (Experimental): Patients randomized to arm A will receive niraparib daily and undergo tumor resection after 28 days (+/- 7 days) of treatment. The participants in both arms will resume/start on treatment with niraparib 2 -4 weeks after surgery . Participants will continue treatment for up to 12 total cycles of treatment or until tumor progression, unacceptable toxicity or withdrawal of consent
  Interventions: Drug: Niraparib; Drug: Resection/Treatment with Niraparib
- Arm B No Treatment with Niraparib (Active Comparator): Subjects in arm B will not receive niraparib prior to surgery. The participants in both arms will resume/start on treatment with niraparib 2 -4 weeks after surgery . Participants will continue treatment for up to 12 total cycles of treatment or until tumor progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Resection/Treatment with Niraparib

INTERVENTIONS:
Drug: Niraparib — Oral, daily, dosage per protocol,4 Weeks
  Other Names: Zejula
  Arms: Arm A Treatment with Niraparib
Drug: Resection/Treatment with Niraparib — The participants in both arms will resume/start on treatment with niraparib 2 -4 weeks after surgery.
  Treatment can be held for an additional 28 days to allow for recovery from surgery, at the investigator's discretion. Participants will continue treatment for up to 12 total cycles of treatment or until tumor progression, unacceptable toxicity or withdrawal of consent.
  Other Names: Zejula

SUMMARY:
This is a randomized, two-arm, open-label, phase 0 trial to assess intratumoral pharmacokinetics and pharmacodynamics of niraparib in subjects with progressive IDH1 or IDH2 mutant glioma.

- This research study involves an experimental treatment called Niraparib.

DETAILED DESCRIPTION:
This is a randomized, two-arm, open-label, phase 0 trial to assess intratumoral pharmacokinetics and pharmacodynamics of niraparib in subjects with progressive IDH1 or IDH2 mutant glioma.

* This research study involves an experimental treatment called Niraparib.
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
* Participants will be randomized into one of two groups

  * Arm A: 1 cycle of Niraparib, followed by surgery, followed by up to 12 cycles of niraparib.
  * Arm B: Surgery followed by up to 12 cycles of niraparib

Participants will receive study treatment for up to 12 Cycles (1 cycle is 28 days long) and will be followed for up to 5 years after the study treatment.

It is expected that about 16 people will take part in this research study.

This research study is a Pilot Study to investigate the study drug's (niraparib) activity in tumor tissue. The U.S. Food and Drug Administration (FDA) has not approved niraparib for this specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age.
* Participants must have histologically or cytologically confirmed glioma, with documented IDH1 and/or IDH2 gene-mutation at time of initial diagnosis
* Participants must have radiographic evidence of progression/recurrence per RANO criteria for low grade gliomas (LGG) on MRI scan
* Participants must be willing and able to get serial MRI scans
* Participants must have surgically accessible tumors and be surgical candidates.
* Participants must be ≥12 weeks from completion of radiation to the CNS.
* Participants must have a baseline brain MRI scan within 21 days prior to Day 1 of treatment.
* Participants must be on a stable or decreasing dose of glucocorticoids for 7 days prior to registration.
* Patient must have Karnofsky Performance Score (KPS) ≥ 70
* Patient must have expected survival of ≥ 6 months.
* Participant must have adequate organ function, defined as follows:

  * Absolute neutrophil count ≥ 1,500/μL
  * Platelets ≥ 100,000/μL
  * Hemoglobin ≥ 9 g/dL
  * Calculated creatinine clearance ≥ 30 mL/min/1.73 m2 using the Cockcroft- Gault equation
  * Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
  * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Patient must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer. (Patients with residual Grade 1 toxicity due to prior chemotherapy or alopecia of any grade are allowed).
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Female participant has a negative urine or serum pregnancy test within 3 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
  * Participant must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

* Participants must have radiographic evidence of primarily disease progression/recurrence per RANO criteria for low grade gliomas (LGG).
* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have had major surgery ≤ 4 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
* Patients may not have received systemic anticancer therapy <28 days prior to their first day of study drug administration. Participants may not have received lomustine < 6 weeks prior to the first day of study drug.
* Patients who received an investigational agent <28 days prior to their first day of study drug administration.
* Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy. Participant must not have received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Participant must not have had diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated).
* Participants who are pregnant or breast-feeding.
* Participants with known hypersensitivity to any of the components of niraparib.
* Participants with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C
* Participants with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate, or participate in the study.
* Participants with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Participants that have had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
* Participant must not have known or symptomatic leptomeningeal metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Drug concentration of niraparib | 1 year
  Drug concentrations of niraparib in enhancing and non-enhancing tumor tissue from subjects treated with the agent for one month prior to surgery.

SECONDARY OUTCOMES:
PARP activity in resected tumors | 1 year
  PARP activity assessed by measuring levels of poly (ADP)-ribose (PAR)s
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0" | Up to one month after discontinuation of treatment
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Median Progression-Free Survival | is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Patients alive without disease progression are censored at date of last disease evaluation up to 5 years
  measured using RANO criteria for low grade glioma
Median Overall Survival | Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive up to 5 years
  calculated with the Kaplan-Meier method and the Log-Rank test will be conducted to compare between the study arms
Duration of Overall Response | one month from start of treatment (Arm A only) and 2, 4, 6 and 12 months out from start of treatment after surgery up to 5 years
  ORR will be calculated as the proportion of patients that are determined to be CR, PR or SD
Response Rate in subjects with recurrent glioma after 1 month of treatment | 1 month
  measured by the Response Assessment in Neuro-Oncology (RANO) Working Group for low-grade gliomas
Response Rate in subjects with residual glioma after surgery | Up to 5 years
  measured by the Response Assessment in Neuro-Oncology (RANO) Working Group for low-grade gliomas (only in patients with subtotal resection)
D-2-hydroxyglutarate (2-HG) levels by MRS | before and one-month post treatment with niraparib up to 3 months
  D-2-hydroxyglutarate (2-HG) levels by MRS
Genomic profile | Up to 5 years
  assessed by whole exome sequencing (WES) performed on resected tumor

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Arrillaga-Romany, MD, Phd, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation